CLINICAL TRIAL: NCT06685705
Title: Comparative Study Between Intrathecal Magnesium Sulfate, Neostigmine and Fentanyl As Adjuvant for Bubivacaine in Postoperative Analgesia in Lower Abdominal Surgeries
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohsen mohamed mohsen mahmoud, Resident at Anesthesia, Intensive Care and Pain Management Department South Egypt cancer Institute, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MgSO4 neostigmine fentanyl
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Magnesium Sulfate; Neostigmine; Fentanyl
Keywords: lower abdominal surgeries
MeSH Terms: interventions — Magnesium Sulfate; Bupivacaine; Neostigmine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: patients will be randomly allocated into one of 3 study designed groups using serial number opaque closed envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- group 1 (Experimental): patients will receive 15 mg of 0.5% hyperbaric bupivacaine + 50 mg Magnesium sulfate intrathecally.
  Interventions: Drug: Magnesium Sulfate and Bupivacaine 0.125%
- group 2 (Experimental): patients will receive 15mg of 0.5% hyperbaric bupivacaine + 50 µg Neostigmine intrathecally
  Interventions: Drug: bupivacaine and Neostigmine
- group3 (Experimental): patients will receive 15mg of 0.5% hyperbaric bupivacaine + 25µg of fentanyl intrathecally.
  Interventions: Drug: fentanyl and bupivacaine

INTERVENTIONS:
Drug: Magnesium Sulfate and Bupivacaine 0.125% — patients will receive 15 mg of 0.5% hyperbaric bupivacaine + 50 mg Magnesium sulfate intrathecally.
  Arms: group 1
Drug: bupivacaine and Neostigmine — patients will receive 15mg of 0.5% hyperbaric bupivacaine + 50 µg Neostigmine intrathecally
  Arms: group 2
Drug: fentanyl and bupivacaine — patients will receive 15mg of 0.5% hyperbaric bupivacaine + 25µg of fentanyl intrathecally.
  Arms: group3

SUMMARY:
Lower abdominal surgeries often result in severe pain, which in turn can cause rapid and shallow breathing, retention of secretions and poor patient compliance. Justifiably, apart from the fear for the surgery outcome, patients are concerned mainly with postoperative pain. If treated inadequately, acute pain can have serious consequences for patient health mainly with postoperative complications, prolonged recovery and increased length of hospital stay. Higher levels of postoperative pain and pain distress are associated with increased morbidity, poorer functional recovery, and reduced quality of life.

Aim of the study To compare the duration, quality of analgesia, and side effects between intrathecal Magnesium sulfate, neostigmine and fentanyl as adjuvant for bubivacaine as postoperative analgesia in lower abdominal surgeries

DETAILED DESCRIPTION:
Effective analgesia aims to minimize patients stress response, pain intensity and distress, and side-effects of large single drug doses (typically an opioid). Numerous analgesic options exist for postoperative analgesia after abdominal surgery, including multiple classes of drugs and routes of administration e.g. parenteral, regional, neuraxial analgesia which include (epidural/intrathecal) techniques, truncal nerve blocks, and systemic drugs infusions.

Spinal anesthesia is a widely used technique in lower abdominal surgeries, offering several benefits such as allowing the patient to remain awake during the procedure, quick onset of action, high success rate, minimal drug dosage, effective sensory and motor blocks, and cost-effectiveness. However, despite these advantages, it can also cause side effects like hypotension, bradycardia, nausea, vomiting, and shivering.

Bupivacaine, is a commonly used local anesthetic, but its use can be limited by the duration of action and potential side effects. To enhance the analgesic effects and prolong the duration of bupivacaine, various adjuvants such as magnesium sulfate, neostigmine, and fentanyl are added intrathecally. Each adjuvant offers unique pharmacological properties that can influence spinal anesthesia's efficacy.

Magnesium sulfate, known for its N-methyl-D-aspartate (NMDA) receptor antagonist properties, decreases sensitivity to both central and peripheral pain stimuli by blocking calcium influx and reducing the excitability of NMDA receptors. Several studies have evaluated the role of magnesium sulfate (MgSO4) as an agent for pain control and reduction of analgesia requirement intra-and post-operatively. In some of these studies, researchers concluded that MgSO4 may reduce the need for opioid analgesic agents.

Neostigmine is a water-soluble, ionized compound that inhibits acetylcholinesterase (AChE). Its indication in FDA is to reverse the effect of non-depolarizing neuromuscular blockers after surgery. The drug is usually administered by intravenous injection, and the main route of excretion is the kidney. Neostigmine should be used with caution in patients with coronary heart disease, arrhythmia, recent acute coronary syndrome and myasthenia gravis. Neostigmine works by preventing the breakdown of the neurotransmitter acetylcholine. Recent studies suggest that this inhibition of acetylcholine degradation strengthens the descending modulation of afferent pain signals, offering a novel method for improving analgesia with minimal dose-related side effects. It enhances spinal cholinergic transmission, potentially increasing the analgesic effects without causing respiratory depression.

Fentanyl, a potent opioid, is commonly used as an adjuvant due to its strong analgesic properties, its primary clinical uses include sedation for intubated patients and managing severe pain, especially in those with renal failure, as it's predominantly metabolized by the liver . Fentanyl is also prescribed for chronic pain patients who have developed a tolerance to other opioids. Fentanyl is more lipid soluble than morphine which is more rapidly eliminated from cerebrospinal fluid. It provides dense blockade with complete intra- and postoperative analgesia without causing hemodynamic instability. It has relatively fewer side effects which are manageable and very well tolerated by the patients.

The comparative effectiveness of these adjuvants in prolonging the duration of analgesia, reducing postoperative opioid requirements, and minimizing adverse effects is crucial for improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* • the American Society of Anesthesiologists (ASA) classification I-II

  * Age >18 up to 55 years old
  * Both sex
  * Patients who will undergo lower abdominal surgeries

Exclusion Criteria:

* • Patients' refusal.

  * Patients with morbid obesity, cardiac diseases, hepatic diseases, renal diseases, diabetes mellitus with polyneuritis.
  * Patients who were in risk-scoring groups American Society of Anesthesia III-IV.
  * Hypertensive patients receiving therapy with adrenergic receptor antagonist, calcium channel blocker and/or angiotensin converting enzyme inhibitor.
  * Patients with coagulation disorders, those receiving any anticoagulants.
  * Any history of allergy to local anesthetic or other drugs used in the study, patients on examining drugs.
  * Any contraindication to spinal anesthesia ( infection at puncture site and increased intracranial tension and Patients with psychiatric illness and neurologic diseases.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
first request of rescue analgesia | baseline
  The time of first request of rescue analgesia calculated from the time of spinal anesthesia.

SECONDARY OUTCOMES:
post operative VAS score | baseline
  post operative VAS score

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Liu W, Bao S, Chen J, Li Y, Gu Y, Ye Q, Hai K. Bupivacaine-fentanyl isobaric spinal anesthesia reduces the risk of ICU admission in elderly patients undergoing lower limb orthopedic surgery. J Orthop Surg Res. 2024 Mar 1;19(1):160. doi: 10.1186/s13018-024-04618-x. PMID 38429736
- [Background] Li LQ, Fang MD, Wang C, Lu HL, Wang LX, Xu HY, Zhang HZ. Comparative evaluation of epidural bupivacaine alone and bupivacaine combined with magnesium sulfate in providing postoperative analgesia: a meta-analysis of randomized controlled trials. BMC Anesthesiol. 2020 Feb 5;20(1):39. doi: 10.1186/s12871-020-0947-8. PMID 32024465
- [Background] Prabhakaraiah UN, Narayanappa AB, Gurulingaswamy S, Kempegowda K, Vijaynagar KA, Hanumantharayappa NB, Ramegowda DS. "Comparison of Nalbuphine Hydrochloride and Fentanyl as an Adjuvant to Bupivacaine for Spinal Anesthesia in Lower Abdominal Surgeries:" A Randomized, Double-blind Study. Anesth Essays Res. 2017 Oct-Dec;11(4):859-863. doi: 10.4103/aer.AER_40_17. PMID 29284839
- [Background] Pandey V, Mohindra BK, Sodhi GS. Comparative evaluation of different doses of intrathecal neostigmine as an adjuvant to bupivacaine for postoperative analgesia. Anesth Essays Res. 2016 Sep-Dec;10(3):538-545. doi: 10.4103/0259-1162.180779. PMID 27746548
- [Background] Si S, Zhao X, Su F, Lu H, Zhang D, Sun L, Wang F, Xu L. New advances in clinical application of neostigmine: no longer focusing solely on increasing skeletal muscle strength. Front Pharmacol. 2023 Aug 4;14:1227496. doi: 10.3389/fphar.2023.1227496. eCollection 2023. PMID 37601044
- [Background] Liao Y, Li Y, Ouyang W. Effects and safety of neostigmine for postoperative recovery of gastrointestinal function: a systematic review and meta-analysis. Ann Palliat Med. 2021 Dec;10(12):12507-12518. doi: 10.21037/apm-21-3291. PMID 35016456
- [Background] Hussien RM, Rabie AH. Sequential intrathecal injection of fentanyl and hyperbaric bupivacaine at different rates: does it make a difference? A randomized controlled trial. Korean J Anesthesiol. 2019 Apr;72(2):150-155. doi: 10.4097/kja.d.18.00173. Epub 2019 Jan 9. PMID 30622224
- [Background] Taher-Baneh N, Ghadamie N, Sarshivi F, Sahraie R, Nasseri K. [Comparison of fentanyl and dexmedetomidine as an adjuvant to bupivacaine for unilateral spinal anesthesia in lower limb surgery: a randomized trial]. Braz J Anesthesiol. 2019 Jul-Aug;69(4):369-376. doi: 10.1016/j.bjan.2019.03.005. Epub 2019 Jul 27. PMID 31362883
- [Background] Pirie K, Traer E, Finniss D, Myles PS, Riedel B. Current approaches to acute postoperative pain management after major abdominal surgery: a narrative review and future directions. Br J Anaesth. 2022 Sep;129(3):378-393. doi: 10.1016/j.bja.2022.05.029. Epub 2022 Jul 6. PMID 35803751